CLINICAL TRIAL: NCT00094237
Title: Subclinical Thyroid Dysfunction and Risk of Myocardial Infarction and Stroke
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1274; R01HL076645 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypothyroidism; Myocardial Infarction; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypothyroidism; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the association of subclinical hypothyroidism and risk of myocardial infarction and stroke in a large prospective cohort of post-menopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease, including myocardial infarction (MI) and stroke, is the leading cause of death for women in the United States. Subclinical hypothyroidism (SCH), in which thyroid hormone levels are in the normal range but thyroid stimulating hormone (TSH) is elevated, has been linked to abnormal lipid profiles, atherosclerosis, and MI. The literature is scant however, and the evidence constrained by small studies, many of cross-sectional design. Both the US Preventive Services Task Force and the Institute of Medicine recently concluded that current data are insufficient to inform clinical decision-making about the need for screening or treatment for SCH.

DESIGN NARRATIVE:

This is a case-cohort study within the 93,676-member Observational Study of the Women's Health Initiative, including 800 women who have experienced an MI, 750 with thrombotic/embolic stroke, and a randomly selected subcohort of 3,200 women density-matched for age, race/ethnicity, and clinical center. Participants have extensive baseline demographic, health, behavioral, and physical exam data and stored serum available. The investigators will measure TSH and thyroid hormone levels in order to identify SCH at entry. Follow-up includes annual health status updates and a physical exam in the third year; >=5 years have passed since enrollment for all women. Thus, using new laboratory studies and existing Women's Health Initiative (WHI) data, they will be able to answer these primary research questions: Among women without a history of thyroid disease, MI, or stroke: 1) Is subclinical hypothyroidism at baseline independently associated with risk of MI? 2) Is subclinical hypothyroidism at baseline independently associated with risk of ischemic stroke? 3) What form of association best describes the relationship between TSH, as a continuous measure, and risk of MI and stroke? 4) What are the population correlates (i.e., race/ethnicity, body mass index (BMI), hormone therapy, comorbidity) of SCH? This information - currently unavailable for middle-aged and older women - is germane to public health and health care policy to define the burden of illness associated with SCH, and to quantify the benefits and costs of eventual population screening and treatment

ELIGIBILITY:
No eligibility criteria

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged 50-79 years, who enrolled in the Women's Health Initiative (WHI) Observational Study (n=93,676). Participants include African American, Asian, Hispanic/Latino and European-American individuals recruited from the communities surrounding the WHI study centers..
Sampling Method: Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hartmann, Principal Investigator — University of North Carolina, Chapel Hill